CLINICAL TRIAL: NCT04047758
Title: Efficacy, Tolerability, and Safety of Palbociclib Combined With an Aromatase Inhibitor in Hormone Receptor-positive/Human Epidermal Growth Factor Receptor 2-negative Locally Advanced Breast Cancer
Brief Title: Palbociclib Combined With an Aromatase Inhibitor in Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Caigang Liu, Director of Department of Breast Surgery, Shengjing Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Shengjing_002
Record Dates: First submitted 2019-08-05; First posted 2019-08-07 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Breast Cancer
Keywords: palbociclib; aromatase inhibitors
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib; Letrozole

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Palbociclib + Letrozole group (Experimental): 210 patients will be randomly assigned to receive treatment with palbociclib and letrozole (palbociclib + letrozole group) .
  Interventions: Drug: Palbociclib + Letrozole
- Letrozole group (Placebo Comparator): 210 patients will be randomly assigned to receive treatment with letrozole (letrozole group).
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Palbociclib + Letrozole — (1) Palbociclib (trade name: Ibrance®; Pfizer Manufacturing Deutschland GmbH, Freiburg, Germany; imported drug license No. H20180040): 125 mg/capsule, 1 capsule by mouth once a day, for 21 successive days, followed by 7 days off treatment [3 weeks on (days 1-21) and 1 week off (days 22-28)], repeated every 28 days. (2) Letrozole (trade name: Femara®; Novartis Pharma Schweiz AG, Switzerland; imported drug license No. H20140149): 2.5 mg/table, 1 table by mouth once a day, continuously for a 28-day cycle.
  Arms: Palbociclib + Letrozole group
Drug: Letrozole — Letrozole (trade name: Femara®; Novartis Pharma Schweiz AG, Switzerland; imported drug license No. H20140149): 2.5 mg/table, 1 table by mouth once a day, continuously for a 28-day cycle.
  Arms: Letrozole group

SUMMARY:
Pfizer's innovative drug palbociclib (trade name: Ibrance®) got China National Drug Administration (CNDA) approval on July 31, 2018. Palbociclib combined with an aromatase inhibitor can be used to treat hormone receptor-positive/human epidermal growth factor receptor 2-negative locally advanced breast cancer or metastatic breast cancer. This brings more treatment options for hormone receptor-positive/human epidermal growth factor receptor 2-negative locally advanced breast cancer. How to scientifically evaluate the efficacy, tolerability, and safety of palbociclib combined with an aromatase inhibitor and to establish a more suitable treatment strategy for Chinese patients is one of the questions that need to be answered in clinical practice. This multi-center parallel-group randomized controlled trial will address on this issue.

DETAILED DESCRIPTION:
Breast cancer is one of the most common cancers in women. Once advanced, it is usually not cured. Studies have shown that patients with advanced breast cancer have a median survival of 2-3 years. For inoperable locally advanced breast cancer, systemic therapy is the first choice of treatment. Systemic treatments of hormone receptor-positive/human epidermal growth factor receptor 2-negative breast cancer mainly include endocrine monotherapy, multi-drug combination therapy and chemotherapy. The overall survival is similar between patients with hormone receptor-positive/human epidermal growth factor receptor 2-negative breast cancer receiving chemotherapy and those receiving endocrine therapy. But quality of life and progression-free survival of patients receiving endocrine therapy are superior to those of receiving chemotherapy. Therefore, both the National Comprehensive Cancer Network (NCCN) and the 2018 Chinese Expert Consensus on the Clinical Diagnosis and Treatment of Advanced Breast Carcinoma guidelines confirm that endocrine therapy is the preferred treatment for hormone receptor-positive/human epidermal growth factor receptor 2-negative breast cancer.

Palbociclib is a cyclin-dependent kinase (CDK) 4/6 inhibitor that reduces the proliferation of estrogen receptor-positive breast cancer cells by blocking cells from the G1 phase to the S phase. Pfizer's innovative drug palbociclib (trade name: Ibrance®) was approved by the China National Drug Administration on July 31, 2018 for the treatment of hormone receptor-positive/human epidermal growth factor receptor 2-negative locally advanced breast cancer or metastatic breast cancer. In addition, aromatase inhibitors such as letrozole (trade name: Femara ®) can prolong the progression-free survival in the first-line therapy for advanced breast cancer to 10-13 months. Palbociclib combined with letrozole has been shown to exhibit stronger inhibitory effects on phosphorylation of retinoblastoma gene (Rt), downstream signaling and tumor growth than monotherapy. Since 2015, palbociclib combined with letrozole has been recommended by the NCCN guideline as one treatment option for advanced breast cancer. However, since palbociclib has been approved for market entry in China for only 1 year, little is reported in China regarding large-sample clinical trials regarding the efficacy, tolerability, and safety of palbociclib combined with an aromatase inhibitor in hormone receptor-positive/human epidermal growth factor receptor 2-negative locally advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histological and imaging findings-confirmed hormone receptor-positive/human epidermal growth factor receptor 2-negative breast cancer;
* postmenopausal patients;
* eligible patients receiving one or more treatment strategies who are followed up in the center where they receive treatment;
* provision of written informed consent.

Exclusion Criteria:

* Age < 18 years;
* pregnant woman;
* participating in other clinical trials.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 24 months
  It is defined as the time from random assignment in a clinical trial to disease progression or death from any cause.

SECONDARY OUTCOMES:
Overall survival | 24 months
  The length of time from either the date of diagnosis or the start of treatment for cancer, that patients diagnosed with the disease are still alive.
Functional Assessment of Cancer Therapy-Breast Cancer (FACT-B) | 24 months
  The FACT-B scale is used for evaluating the survival of patients with breast cancer. The scale consists of 36 items covering physical well-being, social/family well-being, emotional well-being, and functional well-being domains. Higher FACT-B score indicates better heath.
EuroQol five-dimension scale (ED-5Q) | 24 months
  The ED-5Q is a widely used multidimensional measure of health-related quality of life. Higher ED-5Q score indicates better health.

CONTACTS AND LOCATIONS:
Overall Officials: Caigang Liu, Principal Investigator — Shengjing Hospital
Locations (3):
- China (3):
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - Liaoning Provincial People's Hospital, Shenyang, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning